CLINICAL TRIAL: NCT07392450
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Safety, Tolerability, and Efficacy of TAK-755 in Acute Ischemic Stroke
Brief Title: A Study of TAK-755 in Adults With Acute Ischemic Stroke
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-755-2002
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Acute Ischemic Stroke
Keywords: Drug therapy
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part A: TAK-755 (Experimental): Participants will receive a single intravenous (IV) infusion of TAK-755 on Day 1 of Part A. All participants will be followed for up to 90 days post treatment.
  Interventions: Biological: TAK-755
- Part B: TAK-755 (Experimental): Participants will receive a single IV infusion of TAK-755 on Day 1 of Part B. All participants will be followed for up to 90 days post treatment.
  Interventions: Biological: TAK-755
- Part A and B: Placebo (Placebo Comparator): Participants will receive a single IV infusion of TAK-755 matching placebo on Day 1 of Parts A and B. All participants will be followed for up to 90 days post treatment.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: TAK-755 — TAK-755 IV infusion.
  Other Names: rADAMTS13
  Arms: Part A: TAK-755; Part B: TAK-755
Other: Placebo — TAK-755 matching placebo IV infusion.
  Arms: Part A and B: Placebo

SUMMARY:
Acute ischemic stroke (AIS) is a medical emergency that happens because of a sudden stop of blood flow to a part of the brain. This happens when a blood clot forms within the vessel (known as thrombotic occlusion) or a clot originating from somewhere else blocks a blood vessel (known as embolic occlusion). Strokes can cause serious health problems, death, and affect one's quality of life. To reduce long-term damage, it is important to restore blood flow to the brain as soon as possible.

The main aim of this study is to check how safe TAK-755 is, and how well adults with AIS tolerate it. Other aims are to check how well TAK-755 helps participants to manage their everyday activities and to understand whether it helps reduce the seriousness of their stroke symptoms when compared to placebo. A placebo looks like TAK-755, but does not have any medicine in it, to make sure participants do not know which treatment they are taking.

The participants will receive TAK-755 or placebo once; afterwards, their health will be monitored for about 3 months (90 days). All participants, regardless of their assignment to either TAK-755 or placebo, will receive the usual treatment for AIS as per the hospital's normal practice.

ELIGIBILITY:
Inclusion Criteria:

Informed Consent:

1. The participant or legally authorized representative has provided informed consent before the initiation of any trial procedures.

   Age:
2. 18 to 80 years of age, inclusive, at the time of signing the informed consent form.

   Clinical Characteristics:
3. Clinical diagnosis of AIS.
4. Onset of stroke symptoms within 24 hours of enrollment. Wake-up strokes may be included if Last Known Well is within 24 hours of enrollment; time of onset will be considered the time of Last Known Well.
5. National Institutes of Health Stroke Scale score of 6 to 25, indicating moderate to severe stroke.
6. Estimated Modified Rankin Scale score less than (<) 2 prior to AIS presentation, signifying no significant disability.
7. Signs and symptoms consistent with anterior circulation stroke.

   Imaging:
8. Evidence of causative AIS occlusion on imaging (intracranial internal carotid artery [ICA], M1, M2, M3, M4, A1, A2, A3).
9. Evidence of salvageable brain tissue on CT or MR imaging.

Exclusion Criteria:

Medical History:

1. Weight >130 kilograms (kg) or <40 kg.
2. History of severe traumatic brain injury in the past 90 days.
3. History of intracranial hemorrhage.
4. History of intracranial neoplasm except for small meningioma.
5. History of prior stroke in the past 90 days.
6. History of intracranial or intraspinal surgery within the past 90 days.
7. Major surgery or severe trauma in the past 14 days.
8. History of cerebral amyloid angiopathy.
9. History of systemic malignancy, except for locally excised basal cell or squamous cell skin carcinoma with clear margins.
10. Diagnosis of serious, advanced, or terminal illness with anticipated life expectancy of less than 1 year.
11. Participation in other interventional clinical trials within the previous 90 days.
12. Known life-threatening hypersensitivity reaction to TAK-755 or its components.
13. Any prior administration of TAK-755.
14. Administration of caplacizumab in the past 30 days.
15. Administration of von Willebrand factor-containing products in the past 14 days.
16. Baseline conditions (prior to the index AIS event) that prevent an understanding of the nature, scope, and possible consequences of the trial, in the judgment of the investigator.

    Current Stroke Management:
17. Any prior administration (intravenous or intra-arterial) of alteplase or tenecteplase for the index AIS event, as well as any prior administration of prourokinase or reteplase for the index AIS event in countries where approved.
18. Eligible for administration of intravenous thrombolysis (alteplase or tenecteplase, as well as prourokinase or reteplase in countries where approved) for the index AIS event, based on the site's standard clinical guidelines and direct availability.
19. Intent to proceed with endovascular thrombectomy (EVT) for the index AIS event based on eligibility and direct availability.
20. Seizure at time of index AIS event onset.
21. Persistent blood pressure elevation (systolic >=185 millimeters of mercury [mmHg] or diastolic >=110 mm Hg) prior to randomization.
22. Blood glucose <50 milligrams per deciliter (mg/dL) or >400 mg/dL.

    Current Medical Conditions:
23. Active, uncontrolled bleeding.
24. Bleeding diathesis or any other conditions that would pose significant bleeding risk.
25. Inability to undergo MRI or CT.
26. Rapidly improving AIS symptoms.
27. Chronic causative intracranial occlusion.
28. Causative total occlusion of the extracranial ICA.
29. Evidence of septic emboli or bacterial endocarditis.
30. Another clinically significant concomitant disease that may pose additional risks for the participant in the opinion of the investigator.
31. Pregnancy, lactation, or unable to comply with birth control methods or abstinence as specified in the protocol in the opinion of the investigator.

    Imaging:
32. Poor quality imaging that precludes interpretation according to trial protocol.
33. Evidence of significant intracranial mass effect or midline shift.
34. Evidence of occlusion in >1 vascular territory.
35. Evidence of acute or chronic intracranial hemorrhage.
36. Evidence of extensive early ischemic change estimated to be greater than one-third of the middle cerebral artery territory.
37. Evidence of intracranial tumor (except incidental, small meningioma), cerebral aneurysm, or arteriovenous malformation.

    Laboratory:
38. Platelet count <50,000/ cubic millimeters (mm^3).

    Other:
39. Identification by the investigator as being potentially unable or unwilling to cooperate with trial procedures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2027-12-06 (Estimated); Study Completion 2027-12-06 (Estimated)

PRIMARY OUTCOMES:
Part A and B: Percentage of Participants who Develop Symptomatic Intracranial Hemorrhage (sICH) as Defined by the Heidelberg Bleeding Classification System | Up to 120 hours of study drug administration
  The Heidelberg Bleeding Classification System is used to determine whether an Intracranial Hemorrhage (ICH) is symptomatic (sICH) or asymptomatic (aICH). It uses a structured 7-step approach that integrates imaging findings with clinical deterioration. This algorithm includes anatomic description of hemorrhage, adjudication of neurological deterioration, and relatedness between ICH and clinical deterioration. Percentage of participants who develop sICH will be reported.

SECONDARY OUTCOMES:
Part A: Percentage of Participants With Treatment-Related and Unrelated Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | From start of study drug administration up to follow-up (up to 90 days)
  An AE is any untoward medical occurrence in a clinical trial participant, temporally associated with the use of the trial intervention, whether or not the occurrence is considered related to the trial intervention. A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a trial intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the trial intervention or medicinal product. An SAE is defined as any untoward medical occurrence that results in death or is life-threatening or requires inpatient hospitalization or results in significant disability/incapacity or is a congenital anomaly or meets the definitions of other medically significant events. Percentage of participants with TEAEs and SAEs will be reported.
Part A: Percentage of Participants With Severe TEAEs | From start of study drug administration up to follow-up (up to 90 days)
  A TEAE is defined as any event emerging or manifesting at or after the initiation of treatment with a trial intervention or medicinal product or any existing event that worsens in either intensity or frequency following exposure to the trial intervention or medicinal product. A severe TEAE is a type of AE that interrupts usual activities of daily living, or significantly affects clinical status, or may require intensive therapeutic intervention. Percentage of participants with severe TEAEs will be reported.
Part A: Percentage of Participants With Life-Threatening Adverse Events (AEs) | From start of study drug administration up to follow-up (up to 90 days)
  Percentage of participants with life-threatening AEs will be reported.
Part A: Percentage of Participants With AEs of Special Interest (AESIs) | From start of study drug administration up to follow-up (up to 90 days)
  AESIs include sICH, treatment-related aICH, treatment-related extracranial bleeding SAEs, and recurrent AIS. Percentage of participants with AESIs will be reported.
Part A: Percentage of Participants With Clinically Relevant Changes in Vital Signs | From screening up to discharge (up to approximately 8 days)
  Vital signs will include measurement of body temperature, respiratory rate, blood pressure and pulse rate. Any clinically relevant changes in vital signs will be determined at the investigator's discretion.
Part A: Percentage of Participants With Clinically Relevant Changes in Clinical Chemistry and Hematology | From screening up to discharge (up to approximately 8 days)
  Laboratory parameters will include clinical chemistry and hematology. Any clinically relevant changes in laboratory values will be determined at the investigator's discretion.
Part A: Number of Participants With Binding Antibodies to ADAMTS13 | From Day 30 to Day 90
  As per planned analysis, blood sample will be collected to monitor the development of binding and neutralizing antibodies.
Part A: Number of Participants With Neutralizing Antibodies to ADAMTS13 | From Day 30 to Day 90
  As per planned analysis, blood sample will be collected to monitor the development of binding and neutralizing antibodies.
Part A: Percentage of Participants With All-cause Mortality | From start of study drug administration up to follow-up (up to 90 days)
  Percentage of participants who died during the entire study period will be reported.
Part A and B: Percentage of Participants With Modified Rankin Scale (mRS) Score of 0-1 | At Day 90
  The mRS assessment will be used to grade the level of functional independence of participants following a stroke. It is a single-item, global outcome rating scale that categorizes functional independence based on pre-stroke activities, with seven grades representing no (0), no significant (1), slight (2), moderate (3), moderately severe (4), severe (5) disability and death (6). Lower scores indicate better functional outcome. Percentage of participants with mRS of 0-1 will be reported.
Part A and B: Percentage of Participants With mRS Score of 0-2 | At Day 90
  The mRS assessment will be used to grade the level of functional independence of participants following a stroke. It is a single-item, global outcome rating scale that categorizes functional independence based on pre-stroke activities, with seven grades representing no (0), no significant (1), slight (2), moderate (3), moderately severe (4), severe (5) disability and death (6). Lower scores indicate better functional outcome. Percentage of participants with mRS of 0-2 will be reported.
Part A and B: Ordinal Distribution of mRS at Day 90 | At Day 90
  The mRS assessment will be used to grade the level of functional independence of participants following a stroke. It is a single-item, global outcome rating scale that categorizes functional independence based on pre-stroke activities, with seven grades representing no (0), no significant (1), slight (2), moderate (3), moderately severe (4), severe (5) disability and death (6). Lower scores indicate better functional outcome.
Part A and B: Change From Baseline in National Institutes of Health Stroke Scale (NIHSS) Score at 24 Hours | Baseline up to 24 hours
  The NIHSS is a tool to objectively quantify the impairment caused by a stroke. NIHSS assessment is a 15-item impairment scale assessing level of consciousness, extraocular movements, visual fields, facial muscle function, extremity strength, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria), and hemi-inattention (neglect). The total score ranges from 0 to 42 where higher scores indicate greater impairment. A negative change from Baseline indicates improvement.
Part A and B: Percentage of Participants With Recanalization According to Arterial Occlusive Lesion (AOL) Score of 3 | At 24 Hours
  The AOL scale score is a measure of recanalization and ranges from 0 to 3. The grading scale specifically measures the degree of recanalization at the defined target or causative occlusion. A score of 0 is defined as complete occlusion of the target artery. Scores of 1 and 2 account for partial recanalization, with a score of 1 indicating no distal flow while a score of 2 indicates any distal flow. A score of 3 is defined as complete recanalization with any distal flow. Percentage of participants with AOL Score of 3 will be reported.
Part A and B: Percentage of Participants With Reperfusion | At 24 Hours
  Percentage of participants with reperfusion, defined as >90 percent (%) reduction in volume of reversible ischemic tissue (penumbra) from baseline will be reported.
Part A and B: Final Infarct Volume | At 72 Hours
  Final infarct volume at 72 hours or hospital discharge (if earlier than 72 hours) will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/